CLINICAL TRIAL: NCT07136883
Title: Drug-coated Balloon Angioplasty Outcomes After Plain or Scoring Balloon for Vessel Preparation in Patients With Femoropopliteal Arterial Disease. The DASBAD Study: A Prospective Randomized Controlled Trial.
Brief Title: DCB Outcomes After Plain or Scoring Balloon for Vessel Preparation in Patients With Femoropopliteal Arterial Disease
Acronym: DASBAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Sirvent (Other)
Responsible Party: Sponsor-Investigator, Marc Sirvent, Head of Angiology and Vascular Surgery Department, Principal investigator, Hospital de Granollers
Organization: Hospital de Granollers (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-20-080-HGT-CEIMPS
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Femoropopliteal Disease; Drug Coated Balloon; Critical Limb Ischemia (CLI); Peripheral Arterial Disease
Keywords: Periferal Artery Disease; Femoropopliteal Disease; Drug coated balloon; Vessel preparation; randomized controlled trial; Critical Limb Ischemia; scoring balloons; Bailout stent
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POBA (Active Comparator): Vessel preparation using plain old balloon (POBA) prior to using drug coated balloon (Luminor™; Manufacturer: iVascular, S.L.U., Barcelona, Spain) as definitve treatment.
  Interventions: Device: POBA
- Scoring balloon (Active Comparator): Vessel preparation using scoring balloon (AngioSculpt™; Manufacturer: Spectranetics Corporation, Fremont, California, USA) prior to using drug coated balloon (Luminor™; Manufacturer: iVascular, S.L.U., Barcelona, Spain) as definitve treatment.
  Interventions: Device: Scoring Balloon

INTERVENTIONS:
Device: POBA — The intervention consists of preparing the artery with a traditional/regular angioplasty balloon before using the DCB (Luminor™; Manufacturer: iVascular, S.L.U., Barcelona, Spain) as the definitive treatment.
  Other Names: Control group; Group 1
  Arms: POBA
Device: Scoring Balloon — The intervention consists of preparing the artery with a scoring balloon (Angiosculpt™; Manufacturer: Spectranetics Corporation, Fremont, California, USA) before using the DCB (Luminor™; Manufacturer: iVascular, S.L.U., Barcelona, Spain) as the definitive treatment.
  Other Names: Group 2; Treatment group; Intervention group
  Arms: Scoring balloon

SUMMARY:
The goal of this clinical trial is to learn if using a scoring balloon to prepare the femoropopliteal (FP) segment before drug-coated balloon treatment works better than using a regular balloon (called plain old balloon angioplasty, or POBA). This study includes only people with critical limb ischemia (CLI).

The main questions it aims to answer are:

1. Does using a scoring balloon reduce the need for a bailout stent during the procedure?
2. Does a scoring balloon help keep the artery open longer?
3. Is the cost of the scoring balloon procedure similar to the cost of the POBA procedure?

Participants will:

* Receive either a scoring balloon or POBA to prepare the femoropopliteal segment
* Then be treated with a drug-coated balloon in the same segment
* Be monitored during the procedure to see if a bailout stent is needed
* Have follow-up visits to see if the artery remains open

DETAILED DESCRIPTION:
A prospective, single-center clinical trial has been designed with two parallel intervention groups of consecutive CLI patients (Rutherford classification 4-5) with lesions in the F-P segment. It is a single-blind study, where the patient is unaware of their group allocation, but the operator knows the group of each patient.

Patients will be randomly assigned to undergo either conventional balloon angioplasty or AngioSculpt™ scoring balloon angioplasty prior to drug-coated balloon (Luminor™) treatment.

PROCEDURE DESCRIPTION

Antithrombotic Therapy (Pre-, Intra-, and Post-Procedure):

All patients will be on at least single antiplatelet therapy prior to the procedure, receiving either aspirin (100-300 mg/day) or clopidogrel (75 mg/day).

During the procedure, an intravenous bolus of heparin (1 mg/kg body weight) will be administered.

The postprocedural antithrombotic regimen includes:

Clopidogrel: 75 mg/day starting immediately after the index procedure. Aspirin: 100-300 mg/day starting immediately after the index procedure. Dual antiplatelet therapy (DAPT) must be maintained for a minimum of 1 year following the index procedure.

Discontinuation is only permitted if a subsequent procedure requires temporary interruption of one or both antiplatelet agents. In such cases, therapy should be resumed as soon as clinically feasible.

Treatment of Non-Target Lesions:

All significant inflow-limiting lesions (≥50% stenosis) in the study limb must be treated successfully (i.e., ≤30% residual stenosis) prior to initiation of the study index procedure. Treatment should follow the institution's standard of care and reflect current evidence regarding the efficacy of available therapies.

Procedure Sequence of the Target Lesion Treatment:

1. Pre-dilatation of the lesion Pre-dilatation is mandatory and must be performed using either a standard balloon or an AngioSculpt™ scoring balloon, according to the patient's allocation group.

   1. Balloon diameter must match the reference vessel diameter (RVD) in a 1:1 ratio.
   2. The balloon must cover the entire length of the lesion.
   3. A minimum inflation time of 180 seconds is mandatory.
   4. Angiographic imaging must be recorded both before and after pre-dilatation to document the result.
2. Dilatation with Luminor™ drug-coated balloon (DCB) Following pre-dilatation, lesion treatment is completed using the Luminor™ balloon catheter.

   1. A 1:1 RVD to balloon diameter ratio must be used.
   2. The DCB must cover the entire lesion length and extend at least 1 cm proximally and distally beyond the area previously treated with plain balloon angioplasty.
   3. A minimum inflation time of 180 seconds is mandatory.
   4. Angiographic imaging must be recorded post-dilatation to assess the result.

Definition of Procedural Success.

Treatment of the target lesion is considered successful when the final angiographic result meets both of the following criteria:

1. Residual stenosis is <30% by visual estimation, or there is no flow-limiting dissection;
2. Findings are confirmed in two angiographic projections with a minimum angulation difference of 20°.

If the angiographic result is inconclusive, intraoperative duplex ultrasonography must be performed to evaluate lesion patency and result adequacy.

Bail-Out Stenting Criteria:

In cases where the result after DCB angioplasty is inadequate, bail-out stenting is permitted using the following guidelines:

1. Spot stenting should be performed whenever possible.
2. The use of covered stents or drug-coated/drug-eluting stents is not allowed under the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects aged ≥18 years at the time of informed consent. Women of childbearing potential must have a negative pregnancy test within 7 days prior to the procedure and must agree to use a reliable method of contraception during their participation in the study. This requirement does not apply in cases of sterility, infertility, or menopause for at least 12 months.
* Rutherford category 4-5.
* Life expectancy >1 year as assessed by the investigator, based on the patient's medical history.
* Atherosclerotic lesions in the femoropopliteal segment, including in-stent restenosis.
* The subject has been informed, understands the nature of the trial, and has signed the informed consent form to participate in the study. If the subject is capable of understanding and providing informed consent but is physically unable to sign the consent form, an impartial witness may sign on their behalf.
* The patient is willing to comply with all required follow-up visits.
* Presence of at least one patent infragenicular artery (with <50% stenosis) at the end of the procedure.
* Target vessel diameter ≤8 mm.

Exclusion Criteria:

* Pregnant women or women planning to become pregnant during the course of the study.
* Participation in another investigational drug eluting technology study.
* Inability to successfully cross the target lesion with a guidewire (successful crossing is defined as the guidewire tip passing through the lesion without perforation and remaining within the true arterial lumen).
* Inadequate treatment of a proximal lesion (defined as >30% residual stenosis).
* Severe calcification of the target vessel, defined as 270-360 degrees of circumferential calcification (Fanelli grade 4 classification).
* Presence of thrombus in the target vessel.
* Stenosis at the anastomosis site of a bypass.
* Use of atherectomy, thrombectomy, laser, or any similar device in the target lesion/vessel.
* Prior or planned above-ankle amputation of the target limb (this does not apply to transmetatarsal, digital amputations, or ulcer debridement).
* Known coagulopathy, hypercoagulable state, bleeding diathesis, platelet count <80,000/μL or >700,000/μL, or any other hematological disorder.
* History of gastrointestinal bleeding requiring transfusion within the 3 months prior to the study procedure.
* Any subject for whom the use of antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
* Acute coronary syndrome within 30 days prior to the index procedure.
* History of stroke or transient ischemic attack (TIA) within 90 days prior to the index procedure.
* Known hypersensitivity or contraindication to nickel-titanium alloy (Nitinol).
* Other comorbidities that, in the opinion of the investigator, would prevent the subject from receiving this treatment and/or from complying with the follow-up required by this trial.
* Known hypersensitivity or allergy to contrast agents that cannot be managed medically.
* Known hypersensitivity or allergy to heparin, aspirin, paclitaxel, clopidogrel, or other antiplatelet/anticoagulant therapies.
* Contraindication to the use of dual antiplatelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Bailout stenting | At index procedure
  The need for bailout stenting during the index procedure, defined as implantation due to residual stenosis >30% or flow-limiting dissection (type C according to the Kobayashi classification)
Primary patency | 12 months
  Defined by duplex ultrasound as absence of ≥50% restenosis (velocity peak ratio <2.5) and no clinically driven target lesion revascularisation (CD-TLR)

SECONDARY OUTCOMES:
Primary patency | 1, 6, 18 and 24 months
  Defined by duplex ultrasound as absence of ≥50% restenosis (velocity peak ratio <2.5) and no clinically driven target lesion revascularisation (CD-TLR)
Clinically Driven Target Lesion Revascularization (CD-TLR) | At 1 month, every 6 months up to 2 years post-procedure
  Defined as any reintervention due to clinical deterioration*, to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge respectively.
  *defined as a worsening of the patient's quality of life, reflected by the EQ5D-questionnaire, worsening of the Rutherford category with minimal 1 class or worsening of wound healing.
Freedom from device and procedure-related death and freedom from Major Adverse Events (MAE), including Major Adverse Clinical Events (MACE) and Major Adverse Limb Events(MALE) | 1- Freedom from device and procedure-related death through 30 days post-procedure 2- Freedom from MAE (MACE and MALE) at 1 month, every 6 months up to 2 years post-procedure.
  1. Freedom from device and procedure-related death through 30 days post-procedure
  2. Freedom from MAE (MACE and MALE) at 1 month, every 6 months up to 2 years post-procedure.
  Major Adverse Clinical Events (MACE)
  * Death
  * Myocardial infarction
  * Stroke
  * Bleeding complication requiring transfusion
  Freedom from major adverse limb events (MALE) defined as absence of above-the-ankle target limb amputation or major re-intervention to the target lesion(s) (i.e. new bypass graft, jump/interposition graft revision, thrombectomy/thrombolysis, endovascular reintervention…).
Technical success | During the procedure
  Technical success is defined as successful use of a device or technique to re-establish vessel patency with a residual stenosis of <30% by visual estimation and residual stenosis less than 50% by duplex imaging
Procedural success | Occurring <24 hours and <1 month of the procedure
  Procedural success is defined as technical success and completion of the procedure without complications. This represents successful treatment of the vessels (technical success) in the absence of vessel rupture, distal embolization, thrombosis, access complications, and major adverse cardiovascular events.
Wound healing time | The observation period extends from the date of randomization until the earliest of the following: wound healing, death from any cause, or study completion.
  Wound healing time is defined as the number of days required for the wound to achieve complete healing following the index procedure.
Procedural cost | Index procedure
  Procedural cost is defined as the total price in euros of all balloons and stents used

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sirvent, PhD, Principal Investigator — Fundació Privada Hospital Asil de Granollers
Locations (1):
- Fundació Privada Hospital Asil de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data collected within the DASBAD study will be made available to researchers upon reasonable request. Access to the data is controlled to ensure the protection of participant privacy and compliance with applicable data protection laws and regulations. Data will be shared upon revision and approval based on scientific merit by the DASBAD management group (which includes a qualified statistician) of a detailed proposal for their use. The data required for the approved, specified purposes and the trial protocol will be provided after the completion of a data-sharing agreement that will be set up by the principal investigator and his team. All data provided will be anonymized to respect the privacy of patients who have participated in the trial. Estimated timeframe for response will be within 30 days. Requests for data should be addressed to the corresponding author (M.S.G.; msirvent@fphag.org).

REFERENCES:
- [Background] Yu X, Zhang X, Lai Z, Shao J, Zeng R, Ye W, Chen Y, Zhang B, Ma B, Cao W, Liu X, Yuan J, Zheng Y, Yang M, Ye Z, Liu B. One-year outcomes of drug-coated balloon treatment for long femoropopliteal lesions: a multicentre cohort and real-world study. BMC Cardiovasc Disord. 2021 Jul 3;21(1):326. doi: 10.1186/s12872-021-02127-x. PMID 34217209
- [Background] Shishehbor MH, Scheinert D, Jain A, Brodmann M, Tepe G, Ando K, Krishnan P, Iida O, Laird JR, Schneider PA, Rocha-Singh KJ, Zeller T. Comparison of Drug-Coated Balloons vs Bare-Metal Stents in Patients With Femoropopliteal Arterial Disease. J Am Coll Cardiol. 2023 Jan 24;81(3):237-249. doi: 10.1016/j.jacc.2022.10.016. Epub 2022 Nov 1. PMID 36332764
- [Background] Karashima E, Yoda S, Yasuda S, Kajiyama S, Ito H, Kaneko T. Usefulness of the "Non-Slip Element" Percutaneous Transluminal Angioplasty Balloon in the Treatment of Femoropopliteal Arterial Lesions. J Endovasc Ther. 2020 Feb;27(1):102-108. doi: 10.1177/1526602819887954. Epub 2019 Nov 14. PMID 31724469
- [Background] Horie K, Tanaka A, Taguri M, Inoue N. Impact of Scoring Balloons on Percutaneous Transluminal Angioplasty Outcomes in Femoropopliteal Lesions. J Endovasc Ther. 2020 Jun;27(3):481-491. doi: 10.1177/1526602820914618. Epub 2020 Apr 6. PMID 32249658
- [Background] Brodmann M, Lansink W, Guetl K, Micari A, Menk J, Zeller T. Long-Term Outcomes of the 150 mm Drug-Coated Balloon Cohort from the IN.PACT Global Study. Cardiovasc Intervent Radiol. 2022 Sep;45(9):1276-1287. doi: 10.1007/s00270-022-03214-y. Epub 2022 Jul 21. PMID 35864209
- [Background] Tosaka A, Soga Y, Iida O, Ishihara T, Hirano K, Suzuki K, Yokoi H, Nanto S, Nobuyoshi M. Classification and clinical impact of restenosis after femoropopliteal stenting. J Am Coll Cardiol. 2012 Jan 3;59(1):16-23. doi: 10.1016/j.jacc.2011.09.036. PMID 22192663